CLINICAL TRIAL: NCT05678062
Title: Point-of-care Ultrasound Abnormalities in Eclampsia - Prevalence and Association Between Pulmonary Interstitial Syndrome and Cardiac Dysfunction, Brain Natriuretic Peptide, and Serum Albumin
Brief Title: Point-of-care Ultrasound Abnormalities in Eclampsia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cape Town (Other)
Collaborators: Stanford University (Other)
Responsible Party: Principal Investigator, Robert Dyer, Professor Robert Dyer, University of Cape Town
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: POCUS in eclampsia
Record Dates: First submitted 2022-11-22; First posted 2023-01-10 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Eclampsia
Keywords: Pulmonary interstitial syndrome; Cardiac dysfunction; Brain natriuretic peptide
MeSH Terms: conditions — Eclampsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lung- and cardiac ultrasound, as well as optic nerve sheath diameter. (Other): Maternal ultrasound examinations will be performed after normal obstetric treatment protocols have been completed, i.e., the conduction of the study will contribute no delay in routine or emergency patient management. Ultrasound examination will be repeated after 72-96 hours, subject to the same conditions. An ultrasound examination (approximately 35-40 minutes in duration) will be performed. The ultrasound examination will consist of evaluation of lung- and cardiac ultrasound, as well as optic nerve sheath diameter.
  Interventions: Diagnostic Test: Point-of-care ultrasound

INTERVENTIONS:
Diagnostic Test: Point-of-care ultrasound — An ultrasound examination (approximately 35-40 minutes in duration) will be performed. The ultrasound examination will consist of evaluation of lung- and cardiac ultrasound, as well as optic nerve sheath diameter.

SUMMARY:
Preeclampsia (PE) and eclampsia remain leading causes of maternal morbidity and mortality, in both high-, low-and-middle-income countries. Preeclampsia is a complex, multisystem disease which, in its severe form, affects the cardiovascular, renal, hepatic, neurological and haematological systems. Given the complexity of the disease, anaesthesia management for caesarean section in these patients remains challenging. Preeclampsia may be complicated by the development of eclampsia, which involves one or more seizures, which complicates anaesthesia and obstetrics management, and requires. urgent admission and delivery. Recent studies have demonstrated novel markers of severity of PE, including point-of-care ultrasound (POCUS), acid-base changes secondary to low serum albumin, and brain natriuretic peptide (BNP). POCUS is playing an increasing role in perioperative diagnosis, and newer, less expensive devices are continuously being developed. These will in all likelihood play an important role in South Africa in the near future. In a recent trial performed at the University of Cape Town, a comprehensive acid-base analysis in women with PE with severe features demonstrated significant abnormalities in independent acid-base determinants. In addition, strong indications were found that changes in acid-base status following a decrease in serum albumin are more pronounced in early onset PE and may be associated with urgent delivery. In other clinical arenas in critically ill patients, low serum albumin is associated with increased lung water, increased intracranial pressure, and outcome. The research team hypothesised that similar associations might be found in women with late onset preeclampsia with severe features. Using POCUS, it was found that there was no association between serum albumin level and PIS or optic nerve sheath diameter (ONSD). PIS was however associated with cardiac dysfunction, as was BNP.

DETAILED DESCRIPTION:
Preeclampsia is a life-threatening hypertensive disorder involving the heart and vasculature affecting 5-8% of pregnancies. Untreated, 2-10% of women develop eclampsia, defined as new onset of seizures in the setting of preeclampsia. Eclamptic seizures are estimated to occur in 2-8 per 10.000 deliveries in high-income countries (HIC) and with a higher prevalence of up to 16-69 per 10.000 deliveries in low-income countries (LIC). Eclampsia is associated with significant maternal and neonatal morbidity, with a case fatality rate as high as 25-50 % in LIC, and associated with a 16-26 fold odds of death in HIC. Associated maternal complications include intracranial hemorrhage (ICH), cerebral edema, acute kidney injury, acute respiratory syndrome (ARDS), cardiac failure, coagulopathy and postpartum hemorrhage. Obstetric and medical management include seizure prophylaxis and control, aggressive blood pressure management and the urgent delivery of the baby. Anesthesia management can be challenging and has to be tailored to the clinical condition of the eclamptic woman. Unless the usual contraindications to regional anesthesia (RA) apply, spinal anesthesia (SPA) has been described as the method of choice in parturients in whom the Glasgow Coma Scale (GCS) is ≥ 14, and cardiac failure is absent. For patients with persistent decreased level of consciousness, general anesthesia (GA) is recommended. However, in eclamptic women both anesthesia techniques may be associated with significant complications. Raised intracranial pressure (ICP) present in eclamptic women raises the possibility of cerebellar tonsillar herniation in association with SPA. Cardiac diastolic dysfunction, with or without preserved ejection fraction, has been described in preeclamptic women. With preserved ejection fraction, induction of RA or GA is generally hemodynamically well tolerated. However, in women with decreased systolic function, induction of anesthesia can lead to life-threatening cardiovascular collapse, which may only be prevented by cautious titration of anesthesia agents. This might be in conflict with the need to administer high dosages of induction agents to blunt the hypertensive response to tracheal intubation that, if untreated, may lead to life-threatening ICH and pulmonary edema. Consequently, early detection of increased ICP and knowledge of cardiopulmonary function in the individual case are essential to the obstetric anesthetist to guide appropriate management.

Cardiopulmonary and optic nerve sheath point-of-care ultrasound (POCUS) protocols might be particularly suitable for this purpose. These involve a defined bedside ultrasound examination to identify critical cardiopulmonary pathophysiology, which may remain undetected by clinical examination alone. The identification of increased optic nerve sheath diameter (ONSD) on ultrasound may suggest raised ICP.

It is further well documented that the serum brain natriuretic peptide (BNP) level, a marker of cardiac dysfunction, is increased in preeclampsia. However, no data is available to confirm that elevated BNP levels identify those eclamptic women at risk for cardiopulmonary abnormalities.

Therefore, this study is planned to describe the prevalence and severity of cardiac, lung and ONS US abnormalities in women with eclampsia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of preeclampsia following ACOG definition with new onset of tonic-clonic seizures.

Exclusion Criteria:

* Chronic pulmonary disease
* Collagen disorders
* HIV infection if CD4 count <200 cells/ mm3
* Chronic renal or hepatic disease
* Urinary tract infection
* Sepsis
* Body mass index (BMI) > 50 kg/m2
* History of seizure disorder
* Intracranial haemorrhage
* History of benign or malignant intracranial neoplasia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-11-21 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The correlation between pulmonary interstitial syndrome (as identified by lung ultrasound), and cardiac dysfunction on echocardiography, in eclamptic women | 35-40 minutes
  More than 3 B-lines in 2 lung windows bilaterally defines the presence of pulmonary interstitial syndrome. Cardiac dysfunction on echocardiography is defined as raised left ventricular end-diastolic pressure as demonstrated on echocardiography

SECONDARY OUTCOMES:
The correlation between pulmonary interstitial syndrome and optic nerve sheath diameter, serum brain natriuretic peptide and albumin | 35-40 minutes
  Please see description for outcome 1 for pulmonary interstitial syndrome. Abnormal optic nerve sheath diameter is defined as greater than 5.8 mm. Brain natriuretic peptide and serum albumin are continuous variables.
The prevalence of cardiac, lung and optic nerve sheath ultrasound | 35-40 minutes
  Please see definitions as described under Outcome 1 and Outcome 2.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Dyer, MBChB, PhD, Principal Investigator — University of Cape Town
Locations (1):
- Groote Schuur Hospital, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: Yes
The IPD sharing plan is with an Data Transfer Agreement between the two institutions (University of Cape Town and Stanford University), the ultrasound images will be made available to the research team. The results will be shared with fellow clinicians and researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 8 months following publication of results.
Access Criteria: Participants, clinicians and researchers.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-14): https://cdn.clinicaltrials.gov/large-docs/62/NCT05678062/Prot_SAP_000.pdf
  • Informed Consent Form (2022-02-01): https://cdn.clinicaltrials.gov/large-docs/62/NCT05678062/ICF_001.pdf